CLINICAL TRIAL: NCT03269669
Title: Randomized Phase II Trial in Early Relapsing or Refractory Follicular Lymphoma
Brief Title: Obinutuzumab With or Without Umbralisib, Lenalidomide, or Combination Chemotherapy in Treating Patients With Relapsed or Refractory Grade I-IIIa Follicular Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00009; NCI-2017-00009 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1608 (Other: SWOG); S1608 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma; Recurrent Follicular Lymphoma; Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Bendamustine Hydrochloride; Biopsy; Specimen Handling; Cyclophosphamide; Doxorubicin; Lenalidomide; obinutuzumab; Magnetic Resonance Spectroscopy; Prednisone; deltacortene; prednylidene; umbralisib; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (obinutuzumab, umbralisib) (Experimental): CLOSED TO ACCRUAL: Patients receive obinutuzumab IV on day 1 and umbralisib PO daily on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo biopsy and ECHO or MUGA during screening, and PET/CT scans and collection of blood throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Biological: Obinutuzumab; Procedure: Positron Emission Tomography; Drug: Umbralisib
- Arm II (obinutuzumab, lenalidomide) (Experimental): Patients receive obinutuzumab IV on day 1 and lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo biopsy and ECHO or MUGA during screening, and PET/CT scans and collection of blood throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Lenalidomide; Procedure: Multigated Acquisition Scan; Biological: Obinutuzumab; Procedure: Positron Emission Tomography
- Arm III (obinutuzumab, combination chemotherapy) (Active Comparator): PRIOR BENDAMUSTINE-BASED CHEMOTHERAPY: Patients receive obinutuzumab IV on day 1, cyclophosphamide IV on day 1, doxorubicin IV on day 1, vincristine IV on day 1, and prednisone PO on days 1-5. Treatment with obinutuzumab repeats every 21 or 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Treatment with combination chemotherapy repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  PRIOR CHOP CHEMOTHERAPY: Patients receive obinutuzumab IV on day 1, and bendamustine IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for up to 6 or 12 cycles (bendamustine and obinutuzumab, respectively) in the absence of disease progression or unacceptable toxicity.
  Patients undergo biopsy and ECHO or MUGA during screening, and PET/CT scans and collection of blood throughout the trial.
  Interventions: Drug: Bendamustine Hydrochloride; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Biological: Obinutuzumab; Procedure: Positron Emission Tomography; Drug: Prednisone; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Belrapzo; Bendamustin Hydrochloride; Bendeka; CEP 18083; CEP-18083; CEP18083; Cytostasan Hydrochloride; Levact; Ribomustin; SyB L-0501; Treakisym; Treanda; VIVIMUSTA
  Arms: Arm III (obinutuzumab, combination chemotherapy)
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT scans
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Arm III (obinutuzumab, combination chemotherapy)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
  Arms: Arm III (obinutuzumab, combination chemotherapy)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm II (obinutuzumab, lenalidomide)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA 101; GA-101; GA101; Gazyva; huMAB(CD20); R 7159; R-7159; R7159; RO 5072759; RO-5072759; RO5072759
Procedure: Positron Emission Tomography — Undergo PET/CT scans
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Arm III (obinutuzumab, combination chemotherapy)
Drug: Umbralisib — Given PO
  Other Names: 2-((1S)-1-(4-Amino-3-(3-fluoro-4-(1-methylethoxy)phenyl)-1H-pyrazolo(3,4-d)pyrimidin-1-yl)ethyl)-6-fluoro-3-(3-fluorophenyl)-4H-1-benzopyran-4-one; RP-5264; RP5264; TGR 1202; TGR-1202; TGR1202
  Arms: Arm I (obinutuzumab, umbralisib)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Arm III (obinutuzumab, combination chemotherapy)

SUMMARY:
This phase II trial studies how well obinutuzumab with or without umbralisib, lenalidomide, or combination chemotherapy work in treating patients with grade I-IIIa follicular lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Immunotherapy with obinutuzumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Umbralisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as lenalidomide, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Chemotherapy drugs, such as cyclophosphamide, doxorubicin, vincristine, prednisone, and bendamustine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving obinutuzumab with or without umbralisib, lenalidomide, or combination chemotherapy will work better in treating patients with grade I-IIIa follicular lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the complete response rate up to 6 cycles after randomization as defined by centrally read positron emission tomography (PET)/computed tomography (CT) (integral biomarker) of 2 targeted therapeutic regimens (obinutuzumab + umbralisib [TGR-1202] or obinutuzumab + lenalidomide) with obinutuzumab + chemotherapy (cyclophosphamide, doxorubicin hydrochloride [doxorubicin], vincristine sulfate [vincristine], and prednisone [CHOP] or bendamustine hydrochloride [bendamustine]) in patients with early relapsing or refractory follicular lymphoma.

SECONDARY OBJECTIVES:

I. To validate the prognostic association of the m7-FLIPI model, demonstrating that the population of follicular lymphoma patients who respond poorly to chemoimmunotherapy are enriched for having a high-risk m7-FLIPI score, and that the score is associated with progression-free survival (integrated biomarker). (Primary translational medicine) II. To estimate the 30-month sustained complete response rate (CR30) defined by centrally read PET/CT with each of the regimens in this early relapsing or refractory follicular lymphoma population.

III. To estimate best response up to 12 cycles of therapy, progression free survival, duration of response and overall survival with each of the combinations in early relapsing or refractory follicular lymphoma.

IV. To evaluate the adverse effects of each of the regimens in early relapsing or refractory follicular lymphoma.

V. To evaluate the predictive performance of non-invasive genotyping (m7-FLIPI in circulating tumor deoxyribonucleic acid [DNA]) of plasma at study entry relative to standard tumor genotyping (m7-FLIPI) of formalin-fixed paraffin-embedded tumor tissue.

VI. To evaluate the association between the detection of active lymphoma by PET-CT and the detection of circulating tumor DNA in plasma at baseline, after 6 and 12 cycles, and at 30 months after initiation of study therapy.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I (CLOSED TO ACCRUAL): Patients receive obinutuzumab intravenously (IV) on day 1 and umbralisib orally (PO) daily on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive obinutuzumab IV on day 1 and lenalidomide PO on days 1-21. Treatment repeats every 28 days for up 12 cycles in the absence of disease progression or unacceptable toxicity.

ARM III:

PRIOR BENDAMUSTINE-BASED CHEMOTHERAPY: Patients receive obinutuzumab IV on day 1, cyclophosphamide IV on day 1, doxorubicin IV on day 1, vincristine IV on day 1, and prednisone PO on days 1-5. Treatment with obinutuzumab repeats every 21 or 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Treatment with combination chemotherapy repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

PRIOR CHOP CHEMOTHERAPY: Patients receive obinutuzumab IV on day 1 and bendamustine IV over 60 minutes on days 1 and 2. Treatment repeats every 28 days for up to 6 or 12 cycles (bendamustine and obinutuzumab, respectively) in the absence of disease progression or unacceptable toxicity.

Patients in all arms undergo biopsy and echocardiogram (ECHO) or multigated acquisition scan (MUGA) during screening, and PET/CT scans and collection of blood throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have follicular lymphoma (grade I, II or IIIa) confirmed at initial diagnosis and at relapse with identifiable fludeoxyglucose F-18 (FDG) avid disease on PET/CT; patients that have involvement with large cell lymphoma are not eligible
* Patients must have a whole body or limited whole body PET/CT scan performed within 42 days prior to registration
* Patients must have bone marrow biopsy performed within 42 days prior to registration
* Patients must have an indication for therapy as determined by the treating investigator
* All disease must be assessed and documented on the S1608 FDG-PET/CT assessment form
* The intent is to enroll patients with follicular lymphoma (FL) relapsed within 2 years of completing their first course of chemotherapy (CHOP or bendamustine based therapy) + anti-CD20 therapy. Patient is still eligible if he/she received radiation therapy or anti-CD20 therapy prior to chemoimmunotherapy or if maintenance anti-CD20 therapy was administered after chemoimmunotherapy

  * Patients must have either failed to achieve a complete remission, or must have relapsed within 2 years after completing CHOP or bendamustine-containing chemoimmunotherapy (including an anti-CD20 monoclonal antibody), as measured from the last dose of CHOP or bendamustine; relapsed patients must not have received any intervening chemotherapy
  * Patients must have received only 1 course of chemotherapy, containing at least 3 cycles of CHOP or bendamustine; (note that no minimum dose of bendamustine is required)
  * Patients who received any anti-CD20 antibody therapy prior to CHOP or bendamustine are eligible
  * Patients who additionally received any maintenance anti-CD-20 antibody therapy or consolidative radioimmunotherapy within 2 years of the last dose of the CHOP or bendamustine therapy are eligible
  * Involved field or involved site radiation is not considered a line of therapy; examples of eligible prior treatment regimens (note this list is not all inclusive):

    * 1st line rituximab treatment followed years later by bendamustine rituximab
    * Bendamustine rituximab x 4 cycles
    * 1st line rituximab treatment, 2nd line ibritumomab tiuxetan, followed by bendamustine bortezomib rituximab x 6 cycles followed by rituximab maintenance
    * Bendamustine obinutuzumab x 3 cycles
    * CHOP rituximab x 6 cycles followed by rituximab maintenance
* For all forms of systemic therapy, patients must have completed therapy at least 21 days prior to registration; patients must have completed any radioimmunotherapy at least 84 days prior to registration; patients prior treatment related toxicities (except alopecia) must have resolved to grade 1 or less prior to registration
* Patients must have tissue specimens collected prior to registration; patients must be offered participation in biobanking of residual specimens; with patient consent, residuals from the mandatory submission(s) will be banked for future research
* Patients must be >= 18 years of age
* All patients must have a Zubrod performance status of 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1,500/mcL within 28 days prior to registration
* Platelets >= 75,000/mcL within 28 days prior to registration
* Patients must have adequate renal function as documented by a calculated creatinine clearance >= 60 mL/min, within 28 days prior to registration
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (=< 5 x IULN if secondary to lymphoma, Gilbert's syndrome, or medication related [e.g., indinavir, tenofovir, atazanavir]) within 28 days prior to registration
* Direct bilirubin =< 1.5 x IULN (=< 5 x IULN if secondary to lymphoma) within 28 days prior to registration
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x IULN (=< 5 x IULN secondary to lymphoma) within 28 days prior to registration
* Patients must have an echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 42 days prior to registration with a cardiac ejection fraction >= 45%
* Patients with hepatitis B virus infection must have undetectable hepatitis B virus (HBV) on suppressive therapy and no evidence of HBV-related hepatic damage; patients with hepatitis C virus infection are eligible if complete eradication therapy has been successfully completed, and there is no detectable hepatitis C virus (HVC) or related hepatic damage; patients with known human immunodeficiency virus (HIV) infection are eligible if they meet all of the following criteria in addition to the other protocol eligibility criteria:

  * Patient must have no history of acquired immune deficiency syndrome (AIDS)-related complications, other than a history of low CD4+ T-cell count (< 200/mm^3) prior to initiation of combination antiretroviral therapy; on study CD4+ T-cell count may not be informative due to leukemia and should not be used as an exclusion criterion if low
  * Patient must be healthy on the basis of HIV disease with high likelihood of near normal life span were it not for the leukemia
  * Patient must have serum HIV viral load of < 200 copies/mm^3
  * Patient must be on combination antiretroviral therapy with minimal pharmacokinetic interactions with study therapy and minimal overlapping clinical toxicity with protocol therapy; (recommend a regimen of the integrase inhibitor dolutegravir combined with either disoproxil fumarate/emtricitabine or dolutegravir combined with tenofovir alafenamide/emtricitabine)
  * Protease inhibitors and once daily formulations containing cobicistat are NOT allowed due to potential pharmacokinetic interactions with leukemia therapy
  * Stavudine and zidovudine (AZT) are NOT allowed because of overlapping toxicity with protocol therapy
* Patients must be able and willing to receive prophylaxis with daily aspirin, low molecular weight heparin, factor X inhibitors or warfarin if randomized to lenalidomide; patients unable or unwilling to take any listed prophylaxis are NOT eligible
* No second prior malignancy is allowed except for adequately treated basal (or squamous cell) skin cancer, in situ cervical cancer or other cancer for which the patient has been disease free for three years
* Patients must have a complete history and physical examination within 28 days prior to registration
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days and again within 24 hours prior to starting cycle 1 of lenalidomide; further, they must either commit to complete abstinence (true abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence [e.g., calendar, ovulation, symptothermal or post ovulation methods] and withdrawal are not acceptable methods of contraception) from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; while taking lenalidomide, during dose interruptions, and for at least 28 days after the last dose of lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a female who: 1) has achieved menarche at some point; 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure; NOTE: patients not randomized to receive lenalidomide will not be required to undergo serial pregnancy testing or lenalidomide counseling after registration
* Patients must have lactate dehydrogenase (LDH) and beta-2-microglobulin collected within 28 days prior to registration
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Exclusion Criteria:

* Patients must not have clinical evidence of central nervous system involvement by lymphoma since the proposed treatment strategies are not designed to address central nervous system (CNS) involvement adequately; if performed, any laboratory or radiographic tests performed to assess CNS involvement must be negative
* Patients must not have any prior treatment with any PI3K inhibitor, or lenalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2027-01-21 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) | Up to 6 cycles

SECONDARY OUTCOMES:
Sustained complete response rate (CR30) | Up to 30 months
  Defined by centrally read positron emission tomography (PET)/computed tomography (CT).
Progression-free survival (PFS) | From date of registration to date of first observation of progressive disease, or death due to any cause, assessed up to 5 years
  Will be calculated using the method of Kaplan-Meier. 95% confidence for the survival estimates will be constructed using the method of Brookmeyer-Crowley. With 31 eligible patients in each arm, progression free survival at a particular time point, and the 30-month sustained response rate can be estimated to within at least +/- 18% with 95% confidence.
Duration of response (CR, partial response [PR]) | From date of first documentation of response to treatment (CR, PR) to date of first documentation of progression, or death due to any cause, assessed up to 5 years
  Will be calculated using the method of Kaplan-Meier.
Overall survival (OS) | Up to 5 years
  Will be calculated using the method of Kaplan-Meier. 95% confidence for the survival estimates will be constructed using the method of Brookmeyer-Crowley. With 31 eligible patients in each arm, OS at a particular time point, and the 30-month sustained response rate can be estimated to within at least +/- 18% with 95% confidence.
Incidence of adverse events | Up to 5 years
  Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (version 5.0 will be utilized for serious adverse events reporting only). Toxicity rates can be estimated to within at least +/- 18% with 95% confidence.
Non-invasive genotyping and circulating tumor deoxyribonucleic acid (DNA) assessment | Up to 5 years
  Sensitivity, specificity, positive predictive value, negative predictive value, and kappa coefficient will be used to evaluate the concordance. Will evaluate the association of detection of active lymphoma by positron emission tomography-computed tomography and the detection of circulating tumor DNA in plasma at baseline, after 6 and 12 cycles, and at 30 months after initiation of study therapy. Chi-square test will be used to evaluate the association and odds ratio will be calculated
Active lymphoma and circulating tumor DNA in plasma | From baseline up to 30 months after initiation of treatment
  The Cox proportional hazards model will be used to assess the association and odds ratio will be calculated.
m7-FLIPI model validation | Up to 5 years
  The Cox proportional hazards model will be used to assess the association of the m7-FLIPI with to PFS.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Barr, Principal Investigator — SWOG Cancer Research Network
Locations (429):
- United States (429):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - City of Hope Seacliff, Huntington Beach, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - City of Hope Newport Beach, Newport Beach, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Reid Health, Richmond, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin